CLINICAL TRIAL: NCT05854862
Title: Analysis of Relevant Influencing Factors of Glycemic Control in Patients With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20220124-01
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-01

CONDITIONS: Glycemic Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at the analysis of relevant influencing factors of glycemic control in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-90 years with diabetes and the diagnostic criteria of diabetes is according to the World Health Organization in 1999.

Exclusion Criteria:

Patients with stress hyperglycaemia. Patients with severe systemic disease. Patients treated with systemic glucocorticoids within the last three months. Patients without any records about HbA1c, CGM and SMBG.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes who visited in the Department of Endocrinology at the Nanjing First Hospital from August 2013 to the present.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | day 1
  the glycosylated hemoglobin level of patients
TIR | day 1-14
  time in range observed using continuous glucose monitoring

SECONDARY OUTCOMES:
MBG | day 1-14
  mean blood glucose
MAGE | day 1-14
  Mean amplitude of glycemic excursion assessed by continuous glucose monitoring
SD | day 1-14
  the standard deviation of mean glucose
Incidence of hypoglycemia | day 1-14
  Incidence of hypoglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided